CLINICAL TRIAL: NCT04448925
Title: Physiological Responses to Maximal 4-s Sprint Interval Cycling Using Inertial Loading: the Influence of Inter-sprint Recovery Duration
Brief Title: Physiological Responses to Maximal 4-s Sprint Interval Cycling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UTexasAustinHPL
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Exercise, Cardiovascular Function, Fatigue, Muscular Power
MeSH Terms: conditions — Motor Activity; Fatigue

STUDY DESIGN:
Intervention Model Description: Repeated measures, cross-over
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Recovery duration 15 seconds (Experimental): Resting for 15 sec
  Interventions: Other: inertial-load exercise (ILE)
- Recovery duration 30 seconds (Experimental): Resting for 30 sec
  Interventions: Other: inertial-load exercise (ILE)
- Recovery duration 45 seconds (Experimental): Resting for 45 sec
  Interventions: Other: inertial-load exercise (ILE)

INTERVENTIONS:
Other: inertial-load exercise (ILE) — Length of time between exercise bouts

SUMMARY:
The optimal recovery duration depends on the intensity of exercise and in the present study the intensity was maximal power for 4-s while cycling an 'Inertial Load' ergometer (ILE). Recovery duration of 15, 30 and 45-s were given between 30 successive sprints.

DETAILED DESCRIPTION:
All subjects completed an informed consent for this study that was approved by the Institutional Review Board of the University of Texas at Austin.

Study Overview. A randomized, cross-over experimental design was conducted. Each participant visited the laboratory on four occasions which were separated by two to five days. Measurement of body mass, familiarization with experimental procedures and cycling peak oxygen consumption test (VO2peak) were performed on the first visit. Participants took part in inertial-load exercise (ILE) on the remaining test days. On each separate session, a different inter-sprint recovery duration was employed (i.e. 15, 30 or 45-s). Cycling power output, pulmonary gas exchange, vastus lateralis de-oxygenation status, heart rate and blood lactate were measured.

ELIGIBILITY:
Inclusion Criteria:

* healthy participants

Exclusion Criteria:

* unhealthy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
maximal leg power | 10 min

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin Human Performance Laboratory, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
all data will be grouped and averaged

REFERENCES:
- [Derived] Vardarli E, Satiroglu R, Allen JR, Bjellquist-Ledger R, Burton HM, Coyle EF. Physiological responses to maximal 4 s sprint interval cycling using inertial loading: the influence of inter-sprint recovery duration. Eur J Appl Physiol. 2021 Aug;121(8):2295-2304. doi: 10.1007/s00421-021-04677-6. Epub 2021 May 11. PMID 33974126